CLINICAL TRIAL: NCT01902225
Title: A Multicenter Phase I Dose-finding and Preliminary Efficacy Study of the Histone Deacetylase Inhibitor Romidepsin (Istodax®) in Combination With Doxorubicin HCl Liposomal (Doxil®) for the Treatment of Adults With Relapsed or Refractory Cutaneous T-cell Lymphoma
Brief Title: Phase I Dose-finding and Preliminary Efficacy Study of the Istodax® in Combination With Doxil® for the Treatment of Adults With Relapsed or Refractory Cutaneous T-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weiyun Ai (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Weiyun Ai, Clinical Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112516; NCI-2014-01722 (Other: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Lymphoma; T-Cell Lymphoma; Cutaneous Lymphoma
Keywords: Lymphoma; T-Cell; Cutaneous; Doxil; romidepsin; skin
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell; Lymphoma, T-Cell, Cutaneous | interventions — romidepsin; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Istodax, Doxil (Experimental): Istodax; Intravenous; 8-14 mg/m2; Days 1, 8, and 15; over 4 hours
  Doxil; Intravenous; 20 mg/m2; Day 1; over 1 hour
  Interventions: Drug: Istodax; Drug: Doxil

INTERVENTIONS:
Drug: Istodax
  Other Names: Romidepsin
Drug: Doxil
  Other Names: Liposomal doxorubicin

SUMMARY:
This a multi-center, single arm, open-label, Phase I dose-finding and preliminary efficacy study of the combination of the histone deacetylase inhibitor romidepsin (Istodax®) in combination with doxorubicin HCl liposomal (Doxil®) for adult patients with relapsed or refractory cutaneous T-cell lymphoma after at least 2 lines of skin-directed therapy or one prior line of systemic therapy. Patients will be treated with Doxil 20mg/m2 on day 1 and romidepsin 8-14mg/m2 on days 1, 8 and 15, every 28 days, until 2 cycles beyond the best response, 8 cycles, disease progression or intolerability whichever comes first. Importantly, doxil is administered prior to romidepsin on day1 of each cycle. Patients will be followed until disease progression or death whichever comes first.

DETAILED DESCRIPTION:
This a multi-center, single arm, open-label, Phase I dose-finding and preliminary efficacy study of the combination of the histone deacetylase inhibitor romidepsin (Istodax®) in combination with doxorubicin HCl liposomal (Doxil®) for adult patients with relapsed or refractory cutaneous T-cell lymphoma after at least one prior line of systemic therapy.

STUDY ENDPOINTS:

Primary:

MTD will be determined by standard "3+3" dose escalation of romidepsin with a fixed dose of doxorubicin HCl liposomal. Participants will be followed throughout therapy and all adverse events recorded, graded, and given likelihood of relevance to study therapies. Toxicity will be graded by the NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0.

Secondary:

* Response will be assessed by a global response score integrating change in skin disease as measured by the modified severity-weighted assessment tool (mSWAT) score, change in lymph node size, change in visceral disease, and changes in peripheral blood Sézary cells by flow cytometry. CR/PR assignment requires confirmatory assessment in 4 weeks. Skin scores, clinical lymph node, liver and spleen exam, and Sézary cell count assessment will occur on Day 1 of each cycle. Contrasted CT scan of the neck, chest, abdomen and pelvis will be performed at screening for all patients. In patients with lymphadenopathy and/or organomegaly at screening, contrasted CT scans of the neck, chest, abdomen, and pelvis will occur at the end of every third cycle of therapy, within 1 week of cycle 8 completion, and every 6 months for one year after maximal response. All patients will have contrasted CT scans of the neck, chest, abdomen, and pelvis at the time of concern for disease progression in lymph nodes and/or viscera.TTR is the time of the first romidepsin dose to the time of documented objective response (PR/CR). DOR is the time from first objective response (PR or CR) until disease progression.
* TTP will be measured from the time of the first romidepsin dose until disease progression.
* Pruritus will be assessed monthly using a 100 mm visual analog scale. Quality of life will be assessed monthly by Functional Assessment of Cancer Therapy- General (FACT-G), Skindex-29, and ItchyQOL questionnaires.

Exploratory:

Skin lesions will be punch biopsied (two contiguous 5mm biopsies) prior to beginning therapy as standard care of care. Any leftover tissue will be collected for research with consent of patient. Optional single 5mm punch biopsies will be obtained on day 15 of Cycle 2 after infusion of romidepsin, and at disease relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign an informed consent form.
2. Age ≥18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Biopsy-proven, measurable, Stage IB-IVB relapsed or refractory cutaneous T-cell lymphoma after 2 lines of skin-directed therapy or one prior line of systemic therapy (Note: extracorporeal photopheresis will be considered a systemic therapy for this study)
5. All cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study. The only exceptions are participants with erythroderma who have been on corticosteroids for prolonged periods of time (>60 days) without change may continue use of either low dose systemic steroid (equivalent to <10 mg per day of prednisone) or low potency topical steroids are eligible for this study if the frequency and dosage steroids has not changed for 60 days prior to the study. These participants should continue on the same dose of systemic/topical steroid throughout the study period unless they achieve a complete response at which time steroids can be discontinued. Patients are allowed to continue any medications with known activity in T cell lymphomas at the pre-enrollment doses for conditions other than T cell lymphomas (ie, steroids for sarcoidosis) , as long as there is evidence of T cell lymphoma progression while patients were on these agents.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 at study entry.
7. Laboratory test results within these ranges:

   * Absolute neutrophil count ≥750/mm³
   * Platelet count≥75,000/mm³
   * Total bilirubin ≤ 2 x upper limit of normal (ULN)
   * ULN and Aspartate Aminotransferase (ALT) (SGPT) ≤ 3 x ULN.
   * Creatinine < 2 mg/dL
8. Disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast. Patients with early stage of prostate cancer under clinical surveillance without therapy are eligible
9. Negative serum pregnancy test at the time of enrollment for females of childbearing potential.
10. For males and females of child-producing potential, use of effective contraceptive methods during the study to include 2 methods of contraception, one being a condom.
11. Life expectancy >90 days.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females.
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline except topical therapy for mycosis fungoides which must be discontinued 14 days prior to initiation of study therapy.
5. Prior allogeneic hematopoietic cell transplant.
6. Prior solid organ transplant.
7. Cumulative anthracycline exposure greater than 300 mg/m2 doxorubicin equivalents.
8. Known active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of prior hepatitis B virus vaccination are eligible.
9. Central nervous system or meningeal involvement
10. Any known cardiac abnormalities including:

    * Congenital long QT syndrome
    * Baseline QTc interval ≥ 480 milliseconds;
    * Myocardial infarction within 6 months of Cycle 1 Day 1 (C1D1). Subjects with a history of myocardial infarction between 6 and 12 months prior to C1D1 who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event may participate
    * Other significant ECG abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min)
    * Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II- IV. In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present
    * An ECG recorded at screening showing evidence of cardiac ischemia (ST depression of ≥2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present
    * Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions (see Appendix 10) and/or ejection fraction <40% by Multigated Acquisition Scan (MUGA) scan or <50% by echocardiogram and/or MRI
    * A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD)
    * Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes
    * Uncontrolled hypertension, i.e., blood pressure (BP) of ≥160/95; patients with a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria
    * Any cardiac arrhythmia requiring an anti-arrhythmic medication (excluding stable doses of beta-blockers)
    * Any cardiac finding that is deemed ineligible at the discretion of the investigator
11. Patients taking drugs leading to significant QT prolongation and unable to stop drugs prior to treatment
12. Concomitant use of CYP3A4 inhibitors or inducers unless able to stop medication(s) prior to starting study therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03-04 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2020-04-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to 2 years
  The maximum tolerated dose (MTD) will be defined as the highest tested dose level where 33% or more participants experience a dose limiting toxicity (DLT)

SECONDARY OUTCOMES:
Complete response (CR) rate | Up to 2 years
Overall response rate (CR + PR) | Up to 2 years
Time to response (TTR) | Up to 2 years
Duration of response (DOR) | Up to 2 years
Time to progression (TTP) | Up to 2 years
Changes in degree of pruritus | Up to 2 years
Quality of life during therapy | Up to 2 years
Changes in skin related symptoms | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ai Wei, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No